CLINICAL TRIAL: NCT02852967
Title: A Phase 2 Study, Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Efficacy, Tolerability, and Safety of Belumosudil in Subjects With Moderate/Severe Chronic Plaque Psoriasis Who Are Candidates for Systemic Therapy or Phototherapy
Brief Title: A Phase 2, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Belumosudil in Subjects With Moderate/Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KD025-211
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Skin Diseases; Auto-Immune Diseases; Plaque; Dermatology
MeSH Terms: conditions — Skin Diseases; Plaque, Amyloid | interventions — belumosudil; KD025

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Belumosudil 200 mg QD + Placebo (Experimental): One belumosudil 200 mg tablet and 1 matching placebo tablet in the morning and 1 matching placebo tablet in the evening
  Interventions: Drug: Belumosudil; Drug: Placebo
- Belumosudil 200 mg BID (Twice Daily) + Placebo (Experimental): One belumosudil 200 mg tablet and 1 matching placebo tablet in the morning and 1 belumosudil 200 mg tablet in the evening
  Interventions: Drug: Belumosudil; Drug: Placebo
- Belumosudil 400 mg QD + Placebo (Experimental): Two belumosudil 200 mg tablets in the morning and 1 matching placebo tablet in the evening
  Interventions: Drug: Belumosudil; Drug: Placebo
- Belumosudil 600 mg/day (Experimental): Two belumosudil 200 mg tablets in the morning and 1 belumosudil 200 mg tablet in the evening
  Interventions: Drug: Belumosudil
- Placebo (Placebo Comparator): Two matching placebo tablets in the morning and 1 matching placebo tablet in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belumosudil
  Other Names: Rezurock (brand name); KD025
  Arms: Belumosudil 200 mg BID (Twice Daily) + Placebo; Belumosudil 200 mg QD + Placebo; Belumosudil 400 mg QD + Placebo; Belumosudil 600 mg/day
Drug: Placebo — Placebo tablets matching belumosudil
  Arms: Belumosudil 200 mg BID (Twice Daily) + Placebo; Belumosudil 200 mg QD + Placebo; Belumosudil 400 mg QD + Placebo; Placebo

SUMMARY:
This is a phase 2, randomized, placebo-controlled, 2-period study to evaluate the safety, tolerability, and efficacy of belumosudil in adult subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy.

DETAILED DESCRIPTION:
This phase 2, two-period, dose-finding, placebo-controlled study is performed on adult male and female subjects to evaluate the efficacy and safety of subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy.

Period 1: Double-blind, Placebo-controlled Treatment Period

Approximately 110 subjects are planned to be randomly assigned to each of 5 dose cohorts in a 1:1:1:1:1 manner. Each cohort is planned to have 22 subjects who meet eligibility criteria. Subjects are treated with oral (PO) belumosudil tablets or placebo tablets as follows:

* 200 mg belumosudil once daily (QD) (Cohort 1) = one 200 mg belumosudil tablet and 1 matching placebo in the morning and 1 matching placebo in the evening
* 200 mg belumosudil twice daily (BID) (Cohort 2) = one 200 mg belumosudil tablet in the morning and one matching placebo in the morning, and one 200 mg belumosudil tablet in the evening
* 400 mg belumosudil QD (Cohort 3) = two 200 mg belumosudil tablets in the morning and one matching placebo in the evening
* 600 mg/day belumosudil (Cohort 4) = two 200 mg belumosudil tablets in the morning and one 200 mg belumosudil tablet in the evening
* Matching placebo BID (Cohort 5) = 2 matching placebo tablets in the morning and 1 matching placebo tablet in the evening

Subjects in each of the 5 cohorts in Period 1 are treated with study medication for a period of 16 weeks.

Note: Originally, a sample size of 36 subjects per cohort was planned to provide approximately 90% probability ≥ 1 subject in the 5 cohorts would experience an adverse event (AE) that had an underlying rate of ≥ 6% and approximately an 80% probability of ≥ 1 subject in the cohort experiencing an AE that had an underlying rate of ≥ 4%. However, due to a newly available plaque psoriasis treatment, the study is terminated early with 110 subjects.

Period 2: Open-label Treatment Period (with Belumosudil)

All subjects treated for 16 weeks, regardless of treatment with belumosudil (Cohorts 1 through 4) or placebo (Cohort 5) are given the option to receive 400 mg belumosudil QD for an additional 32 weeks (Week 16 through Week 48).

Follow-up Period

All subjects have a safety evaluation 30 days after the last dose of study drug.

Efficacy is assessed by the following scores at scheduled time points throughout the study:

* Psoriasis Area and Severity Index (PASI): Measure of psoriasis disease severity using average redness, thickness, and scaliness of lesions (each lesion graded 0 to 4), combined into single score ranging on a scale from 0 (no disease) to 72 (maximum disease)
* Physician's Global Assessment (PGA): Physician's assessment of a subject's psoriasis, relative to baseline, ranging on a scale from 1 (100% clearing of psoriasis) to 6 (poor to no clearing)
* Dermatology Life Quality Index (DLQI): Skin disease-specific instrument for assessing impact of disease on subject's quality of life ranging on a scale from 0 (no effect on subject's life) to 30 (extremely large effect on subject's life)

Safety is assessed by;

* AEs and serious AE (SAEs)
* Physical examination
* Vital sign measurements
* Clinical laboratory evaluations
* Electrocardiogram
* Reasons for discontinuation due to toxicity analyses

The maximum duration for subjects who complete Period 1 (Double-blind, Placebo-controlled) is 24 weeks (up to 4-week Screening, 16-week Period 1 treatment, and 4-week Follow-up). The maximum duration for subjects who complete Period 2 (Open-label) is 56 weeks (up to 4-week Screening, 16-week Double-blind Treatment Period, 32-week Open-label Treatment Period, and 4-week Follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects between the ages of 18 and 65 years
* Able to provide written Informed Consent Form prior to the performance of any study-specific procedures
* Diagnosis of moderate to severe chronic plaque psoriasis and a candidate for systemic therapy or phototherapy
* PASI of ≥ 12 at screening and prior to the first dose of study drug, confirmed at Week 1 Day 1 (Baseline)
* ≥ 10% PASI body surface area involvement at screening and prior to the first dose of study drug, confirmed at Baseline
* Willing to avoid tanning devices
* Adequate bone marrow function:

  * Absolute neutrophil count > 1500/mm^3
  * Hemoglobin > 9.0 g/dL
  * Platelets > 100,000/mm^3
* Adequate safety laboratory values:

  * Serum total bilirubin within normal limits (WNL)
  * Aspartate aminotransferase (AST) and alalnine aminotransferase (ALT) < 2 × upper limit of normal (ULN)
  * Serum creatinine < 1.5 × ULN
* Female subjects of childbearing potential with a negative pregnancy test at screening. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who had any evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to prior chemotherapy, antiestrogens, or ovarian suppression

  * Women of childbearing potential (i.e., menstruating women) had to have a negative urine pregnancy test (positive urine tests were to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug
  * Sexually active women of childbearing potential enrolled in the study had to agree to use 2 forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control included: (a) intrauterine device plus 1 barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; and (c) 2 barrier methods. Effective barrier methods were male or female condoms, diaphragms, and spermicides (creams or gels that contained a chemical to kill sperm); or (d) a vasectomized partner
* For male patients who were sexually active and who were partners of premenopausal women: agreed to use 2 forms of contraception as defined above during the treatment period and for at least 3 months after the last dose of study drug
* Willing to complete all study measurements and assessments in compliance with the protocol

Exclusion Criteria:

* Non-plaque or drug-induced (antimalarials, lithium) psoriasis (If subject was taking angiotensin II receptor blockers or beta blockers doses must have been stable for 6 months prior to study entry)
* Used systemic corticosteroids within 12 weeks prior to study entry
* Used topical corticosteroids except to the face, groin, or scalp
* Used methotrexate, retinoids (such as acitretin), or calcineurin inhibitors (such as cyclosporine) within 4 weeks prior to study entry
* Phototherapy within 4 weeks prior to study entry
* Biologic therapies, including antibodies to IL-17; anti-tumor necrosis factor-alpha; and anti-IL-12 & IL-23 within 3 months prior to study entry
* Current use of an inhibitor or inducer of CYP3A4
* Active viral, fungal, or bacterial skin infection (other than nail fungal infection).
* Pregnant or lactating woman
* History of gastrointestinal (GI) surgery including any bariatric surgery, or any GI condition that might interfere with drug absorption
* Participating in another study with an investigational drug or within 28 days or 5 half-lives of the investigational drug (whichever was longer) of study entry
* History or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the investigator, unsuitable for the study
* Regular and/or excessive use of alcohol within 2 years prior to study entry defined as alcohol intake > 14 drinks per week in a man or > 7 drinks per week in a woman. Approximately 10 g of alcohol equaled one "drink" unit. One unit equaled 1 ounce of distilled spirits, one 12-ounce beer, or one 4-ounce glass of wine
* QT interval data corrected using Fridericia's formula (QTcF) > 450 msec (average of 3 readings) during screening
* Exposure to belumosudil or known allergy/sensitivity to belumosudil within the last 6 months prior to study entry or any other ROCK-2 inhibitor
* History or presence of any of the following:

  * ALT or AST > 2.0 × ULN at screening
  * Renal disease and/or serum creatinine > 1.5 × ULN at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - University of California, Irvine - Dermatology Clinical Research Center, Irvine, California
  - Dermatology Research Associates, Los Angeles, California
  - Renstar Medical Research, Ocala, Florida
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Dermatology Specialists Research, New Albany, Indiana
  - Dermatology Specialists Research, Louisville, Kentucky
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Sadick Research Group, New York, New York
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Suzanne Bruce and Associates, Katy, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Belumosudil 200 mg QD + Placebo: One belumosudil 200 mg tablet and 1 matching placebo tablet in the morning and 1 matching placebo tablet in the evening
  Belumosudil: Belumosudil tablets
  Placebo: Placebo tablets matching belumosudil
- Belumosudil 200 mg BID (Twice Daily) + Placebo: One belumosudil 200 mg tablet and 1 matching placebo tablet in the morning and 1 belumosudil 200 mg tablet in the evening
  Belumosudil: Belumosudil tablets
  Placebo: Placebo tablets matching belumosudil
- Belumosudil 400 mg QD + Placebo: Two belumosudil 200 mg tablets in the morning and 1 matching placebo tablet in the evening
  Belumosudil: Belumosudil tablets
  Placebo: Placebo tablets matching belumosudil
- Belumosudil 600 mg/Day: Two belumosudil 200 mg tablets in the morning and 1 belumosudil 200 mg tablet in the evening
  Belumosudil: Belumosudil tablets
Period: Overall Study
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo
Started | 23 | 22 | 21 | 26 | 18
Completed Period 1: Double-blind | 14 | 15 | 17 | 16 | 10
Completed Period 2: Open-label | 11 | 8 | 13 | 11 | 14
Completed | 9 | 6 | 9 | 4 | 2
Not Completed | 14 | 16 | 12 | 22 | 16
Not completed — Adverse Event | 3 | 1 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 3 | 4 | 4
Not completed — Withdrawal by Subject | 6 | 12 | 7 | 10 | 10
Not completed — SAE | 0 | 0 | 0 | 3 | 0
Not completed — Elevated Liver Enzymes | 2 | 0 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 1 | 1 | 0
Not completed — Dispensing Drug Violation | 0 | 0 | 1 | 0 | 0
Not completed — Inclusion/Exclusion Violation | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | Total
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (8.9) | 46.2 (9.6) | 43.0 (11.4) | 43.5 (11.5) | 45.7 (14.2) | 45.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 14 | 15 | 11 | 69
  Male | 7 | 9 | 7 | 11 | 7 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 4 | 8 | 2 | 23
  Not Hispanic or Latino | 18 | 18 | 16 | 18 | 15 | 85
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 1 | 2 | 1 | 3 | 8
  White | 20 | 19 | 17 | 24 | 14 | 94
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2
BMI (Mean) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 33.8 (9.9) | 30.7 (7.0) | 29.9 (7.4) | 33.1 (10.7) | 32 (6.7) | 32.0 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percentage of Subjects With a ≥ 75% Decrease in PASI (PASI 75) at Week 16 (Double-blind Period)--LOCF and Observed
Description: The percentage of subjects who exhibited a 75% decrease or greater in the Psoriasis Area and Severity Index Score (PASI 75) whether they completed 16 weeks of treatment or not (last observation carried forward [LOCF]) and those who did complete 16 weeks of treatment (observed).
  [PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 16 weeks
Population: PASI 75 determined by Last Observation Carried Forward (LOCF) and Observed at the end of Double-blind Period: 16 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Belumosudil: All subjects in the Belumosudil 200 mg QD, 200 mg BID, 400 mg QD, and 600 mg/day cohorts
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Percentage of participants
  LOCF (%) | 8.7 [1.1 to 28.0] | 9.1 [1.1 to 29.2] | 19.0 [5.4 to 41.9] | 7.7 [0.9 to 25.1] | 16.7 [3.6 to 41.4] | 10.9 [5.3 to 19.1]
  Observed (%): number analyzed (Participants) | 14 | 15 | 17 | 16 | 10 | 62
  Observed (%) | 7.1 [0.2 to 33.9] | 13.3 [1.7 to 40.5] | 23.5 [6.8 to 49.9] | 12.5 [1.6 to 38.3] | 30.0 [6.7 to 65.2] | 14.5 [6.9 to 25.8]
Statistical Analysis 1: Comparison: Belumosudil 200 mg QD + Placebo; LOCF at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 200 mg QD + placebo (n = 23) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 18) who achieved PASI 75; Test type: Superiority; p = 0.6384, Fisher Exact
Statistical Analysis 2: Comparison: Belumosudil 200 mg BID (Twice Daily) + Placebo; LOCF at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 200 mg BID + placebo (n = 22) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 18) who achieved PASI 75; Test type: Superiority; p = 0.6419, Fisher Exact
Statistical Analysis 3: Comparison: Belumosudil 400 mg QD + Placebo; LOCF at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 400 mg QD + placebo (n = 21) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 18) who achieved PASI 75; Test type: Superiority; p > 0.9999, Fisher Exact
Statistical Analysis 4: Comparison: Belumosudil 600 mg/Day; LOCF at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 600 mg (n = 26) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 18) who achieved PASI 75; Test type: Superiority; p = 0.3859, Fisher Exact
Statistical Analysis 5: Comparison: All Belumosudil; LOCF at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of all subjects treated with belumosudil (n = 92) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 18) who achieved PASI 75; Test type: Superiority; p = 0.4435, Fisher Exact
Statistical Analysis 6: Comparison: Belumosudil 200 mg QD + Placebo; Observed at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 200 mg QD + placebo (n = 14) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 10) who achieved PASI 75; Test type: Superiority; p = 0.2721, Fisher Exact
Statistical Analysis 7: Comparison: Belumosudil 200 mg BID (Twice Daily) + Placebo; Observed at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 200 mg BID+ Placebo (n = 15) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 10) who achieved PASI 75; Test type: Superiority; p = 0.3577, Fisher Exact
Statistical Analysis 8: Comparison: Belumosudil 400 mg QD + Placebo; Observed at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 500 mg QD + Placebo (n = 17) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 10) who achieved PASI 75; Test type: Superiority; p > 0.9999, Fisher Exact
Statistical Analysis 9: Comparison: Belumosudil 600 mg/Day; Observed at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of subjects treated with belumosudil 600 mg/day (n = 16) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 10) who achieved PASI 75; Test type: Superiority; p = 0.3402, Fisher Exact
Statistical Analysis 10: Comparison: All Belumosudil; Observed at 16 weeks (Double-blind Treatment Period): Fisher's Exact Method analysis of the percentage of all subjects treated with belumosudil 200 mg QD + Placebo (n = 62) who achieved PASI 75 compared to the percentage of subjects treated with placebo (n = 10) who achieved PASI 75; Test type: Superiority; p = 0.3542, Fisher Exact

2. Secondary Outcome: Efficacy: Mean Change of Raw PASI Score From Baseline to Week 16 and Week 48--LOCF and Observed
Description: The mean change in the raw Psoriasis Area and Severity Index (PASI) score from baseline score to Week 16 and to Week 48 whether the subject completed 16 and 48 weeks, respectively (last observation carried forward [LOCF]), or for only those subjects who completed 16 and 48 weeks (observed), respectively. Negative values represent favorable results; positive values represent unfavorable results.
  [The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 48 weeks
Population: Not all subjects had PASI performed
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Score on a scale
  Baseline | 18.93 (8.31) | 20.60 (8.27) | 18.82 (6.08) | 19.80 (9.03) | 20.72 (8.08) | 19.55 (7.97)
  Change at Week 16--LOCF: number analyzed (Participants) | 23 | 21 | 20 | 24 | 17 | 88
  Change at Week 16--LOCF | -5.69 (8.59) | -4.49 (7.44) | -5.0 (8.31) | -4.63 (8.04) | -5.68 (12.31) | -4.96 (7.98)
  Change at Week 16--Observed: number analyzed (Participants) | 14 | 15 | 17 | 16 | 10 | 62
  Change at Week 16--Observed | -3.75 (8.62) | -6.29 (6.45) | -4.96 (8.72) | -3.81 (5.37) | -8.44 (15.36) | -4.71 (7.31)
  Change at Week 48--LOCF: number analyzed (Participants) | 14 | 12 | 16 | 14 | 10 | 56
  Change at Week 48--LOCF | -3.85 (10.53) | -6.38 (5.16) | -9.01 (7.63) | -0.83 (7.73) | -9.56 (18.98) | -5.11 (8.45)
  Change at Week 48--Observed: number analyzed (Participants) | 10 | 5 | 9 | 3 | 2 | 27
  Change at Week 48--Observed | -5.93 (11.26) | -5.30 (5.88) | -12.99 (6.71) | -4.27 (2.16) | 9.45 (21.00) | -7.98 (8.76)

3. Secondary Outcome: Efficacy: Percentage Change in Mean PASI Score From Baseline to Week 16 and to Week 48--LOCF and Observed
Description: The percentage (%) change in the mean Psoriasis Area and Severity Index (PASI) score from baseline ore to Week 16 and to Week 48 whether the subject completed 16 and 48 weeks, respectively (last observation carried forward [LOCF]) or for only those subjects who completed 16 and 48 weeks (observed), respectively.
  [The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 48 weeks
Population: Not all subjects had PASI performed
Measure: Mean (Standard Deviation); unit: Percentage Change in PASI Score
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Percentage Change in PASI Score
  Change (%) at Week 16--LOCF: number analyzed (Participants) | 23 | 21 | 20 | 24 | 17 | 88
  Change (%) at Week 16--LOCF | -27.17 (37.60) | -19.61 (35.60) | -24.31 (42.74) | -20.07 (31.20) | -18.23 (43.93) | -22.78 (36.27)
  Change (%) at Week 16--Observed: number analyzed (Participants) | 14 | 15 | 17 | 16 | 10 | 62
  Change (%) at Week 16--Observed | -15.21 (36.90) | -29.70 (30.72) | -24.17 (44.61) | -20.22 (30.16) | -25.09 (54.31) | -22.46 (35.77)
  Change (%) at Week 48--LOCF: number analyzed (Participants) | 14 | 12 | 16 | 14 | 10 | 56
  Change (%) at Week 48--LOCF | -12.82 (40.33) | -30.75 (24.51) | -46.97 (39.90) | -9.31 (41.28) | -19.89 (90.61) | -25.54 (39.87)
  Change (%) at Week 48--Observed: number analyzed (Participants) | 10 | 5 | 9 | 3 | 2 | 27
  Change (%) at Week 48--Observed | -21.81 (38.75) | -30.02 (34.39) | -63.04 (29.04) | -33.16 (15.48) | 84.98 (166.19) | -38.33 (36.22)

4. Secondary Outcome: Efficacy: Number of Subjects With Clear or Almost Clear PGA at Week 16--LOCF
Description: The number of subjects who had a "Clear" or "Almost Clear" assessment, using the Physician Global Assessment Scale (PGA), at Week 16 of all subjects whether they completed 16 weeks or not (last observation carried forward [LOCF]) [The PGA documents the physician's assessment of the subject's psoriasis and was assessed relative to baseline conditions. The PGA rating is from 1-6, where 1 = 100% clearing of psoriasis (clear), 5 = 0 to 24% clearing (little or no change), and 6 = worse.]
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Participants | 1 | 0 | 2 | 1 | 2 | 4

5. Secondary Outcome: Efficacy: Percentage of Subjects With Clear or Almost Clear PGA Comparing Belumosudil to Placebo at Week 16--LOCF
Description: The percentage (%) of subjects who had a "Clear" or "Almost Clear" assessment using the Physician Global Assessment Scale at Week 16 of belumosudil vs. placebo for all subjects whether they completed 16 weeks or not (last observation carried forward [LOCF]).
  [The PGA documents the physician's assessment of the subject's psoriasis and was assessed relative to baseline conditions. The PGA rating is from 1-6, where 1 = 100% clearing of psoriasis (clear), 5 = 0 to 24% clearing (little or no change), and 6 = worse.]
Time Frame: 16 weeks
Population: Not all subjects had a response to treatment
Measure: Number (95% Confidence Interval); unit: Percentage (%) of subjects
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 92
Percentage (%) of subjects | -6.8 [-23.5 to 10.0] | -11.1 [-25.6 to 3.4] | -1.6 [-20.8 to 17.6] | -7.3 [-23.6 to 9.0] | -6.8 [-21.9 to 8.3]
Statistical Analysis 1: Comparison: Belumosudil 200 mg QD + Placebo; Percentage of subjects treated with belumosudil compared to placebo who had a PGA rating of clear or almost clear; Test type: Superiority; p = 0.5728, Fisher Exact
Statistical Analysis 2: Comparison: Belumosudil 200 mg BID (Twice Daily) + Placebo; Percentage of subjects treated with belumosudil compared to placebo who had a PGA rating of clear or almost clear; Test type: Superiority; p = 0.1962, Fisher Exact
Statistical Analysis 3: Comparison: Belumosudil 400 mg QD + Placebo; Test type: Superiority — Percentage of subjects treated with belumosudil compared to placebo who had a PGA rating of clear or almost clear; p > 0.9999, Fisher Exact
Statistical Analysis 4: Comparison: Belumosudil 600 mg/Day; Percentage of subjects treated with belumosudil compared to placebo who had a PGA rating of clear or almost clear; Test type: Superiority; p = 0.5583, Fisher Exact
Statistical Analysis 5: Comparison: All Belumosudil; Percentage of subjects treated with belumosudil compared to placebo who had a PGA rating of clear or almost clear; Test type: Superiority; p = 0.2538, Fisher Exact

6. Secondary Outcome: Efficacy: Change in Mean DLQI Raw Score at Week 16 and at Week 48
Description: Changes in mean Dermatology Life Quality Index (DLQI) score from baseline at Week 16 (End of Double-blind Period) and at Week 48 (End of Study Treatment).
  [The DLQI is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life. DLQI scoring as measured on subject's life: 0-1 = no effect; 2-5 = small effect; 6-10 = moderate effect; 11 to 20 = very large effect; 21 to 30 = extremely large effect. Change < 0% is improvement; > 0% is worsening. The total rating ranges from 0 (no effect on a subject's life) to 30 (extremely large effect on a subject's life.]
Time Frame: Up to 48 weeks
Population: Not all subjects could be evaluated at all visits.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Score on a scale
  Baseline | 10.6 (6.3) | 16.5 (9.4) | 12.2 (6.5) | 11.0 (7.1) | 10.3 (6.4) | 12.5 (7.7)
  Change at Week 16: number analyzed (Participants) | 14 | 15 | 17 | 16 | 10 | 62
  Change at Week 16 | -2.2 (5.6) | -3.4 (4.0) | -2.5 (6.0) | -2.3 (7.0) | -4.0 (6.7) | -2.6 (5.7)
  Change at Week 48: number analyzed (Participants) | 10 | 5 | 9 | 3 | 2 | 27
  Change at Week 48 | -6.5 (5.1) | -1.0 (8.6) | -5.2 (6.9) | -3.7 (3.2) | -3.0 (2.8) | -4.7 (6.3)

7. Secondary Outcome: Efficacy: Percentage Change of Mean DLQI Score From Baseline to Week 16 and Week 48
Description: Mean percentage changes in Dermatology Life Quality Index (DLQI) from baseline at Week 16 (End of Double-blind Period) and at Week 48 (End of Study Treatment).
  [The DLQI is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life. The rating ranges from 0 (no effect on a subject's life) to 30 (extremely large effect on a subject's life.]
Time Frame: Up to 48 weeks
Population: Not all subjects could be evaluated at all visits. Mean decrease in mean DLQI score is favorable; mean increase is not favorable
Measure: Mean (Standard Deviation); unit: Percentage change of DLQI score
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Percentage change of DLQI score
  Percentage Change at Week 16: number analyzed (Participants) | 14 | 14 | 17 | 15 | 10 | 60
  Percentage Change at Week 16 | -5.73 (60.75) | -14.8 (28.78) | -22.22 (48.60) | -6.4 (79.95) | -40.30 (47.83) | -12.55 (56.58)
  Percentage Change at Week 48: number analyzed (Participants) | 10 | 4 | 9 | 2 | 2 | 25
  Percentage Change at Week 48 | -32.41 (86.97) | 3.54 (54.32) | -45.60 (45.84) | -53.73 (45.24) | -54.17 (41.25) | -33.11 (65.64)

8. Secondary Outcome: Safety: Number of Subjects With TEAEs, SAEs, and Deaths Throughout the Study
Description: The number of subjects who had treatment-emergent adverse events (TEAEs), severity of TEAEs, relationship of TEAEs to study medication, serious TEAEs (SAEs), dose interruption, discontinuations, and deaths.
  Treatment-emergent adverse events (TEAEs) are AEs that are not present before the first dose of IMP or that are present before the first dose of IMP but worsen in intensity during exposure to IMP.
  Severity: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = Death. Related to study medication is defined as possible related, probable related, and related
Time Frame: Approximately 52 weeks: up to 48 weeks of treatment and 30-day follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Belumosudil 200 mg QD + Placebo: One belumosudil 200 mg tablet and 1 matching placebo tablet in the morning and 1 matching placebo tablet in the evening
  Belumosudil
  Placebo: Placebo tablets matching belumosudil
- Belumosudil 200 mg BID (Twice Daily) + Placebo: One belumosudil 200 mg tablet and 1 matching placebo tablet in the morning and 1 belumosudil 200 mg tablet in the evening
  Belumosudil
  Placebo: Placebo tablets matching belumosudil
- Belumosudil 400 mg QD + Placebo: Two belumosudil 200 mg tablets in the morning and 1 matching placebo tablet in the evening
  Belumosudil
  Placebo: Placebo tablets matching belumosudil
- Belumosudil 600 mg/Day: Two belumosudil 200 mg tablets in the morning and 1 belumosudil 200 mg tablet in the evening
  Belumosudil
- All Belumosudile: All subjects from all cohorts who received belumosudil
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudile
Number analyzed (Participants) | 23 | 22 | 21 | 26 | 18 | 92
Participants
  At least 1 TEAE | 14 | 13 | 14 | 16 | 11 | 57
  Grade 3 or Greater TEAE | 2 | 3 | 0 | 5 | 2 | 10
  Related TEAE | 8 | 6 | 5 | 9 | 6 | 28
  Related Grade 3 or Greater TEAE | 1 | 1 | 0 | 3 | 1 | 5
  Leading to Dose Interruption | 1 | 1 | 1 | 4 | 0 | 7
  SAE | 1 | 0 | 0 | 3 | 1 | 4
  Related SAE | 0 | 0 | 0 | 0 | 0 | 0
  Leading to Discontinuation | 6 | 1 | 1 | 7 | 3 | 15
  Deaths | 1 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Approximately 52 weeks: up to 48 weeks of treatment and 30-day follow-up
Description: Adverse events were categorized as treatment-emergent adverse events (TEAEs). TEAEs are AEs that are not present before the first dose of IMP or that are present before the first dose of IMP but worsen in intensity during exposure to IMP.
Groups:
- All Belumosudil: All subjects from all cohorts who received belumosudil
Arm/Group | Belumosudil 200 mg QD + Placebo | Belumosudil 200 mg BID (Twice Daily) + Placebo | Belumosudil 400 mg QD + Placebo | Belumosudil 600 mg/Day | Placebo | All Belumosudil
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/22 | 0/21 | 0/26 | 0/18 | 1/92
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/22 | 0/21 | 3/26 | 1/18 | 1/92
Other Adverse Events (participants affected / at risk) | 14/23 | 13/22 | 14/21 | 16/26 | 11/92 | 57/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil 200 mg QD + Placebo (N=23) | Belumosudil 200 mg BID (Twice Daily) + Placebo (N=22) | Belumosudil 400 mg QD + Placebo (N=21) | Belumosudil 600 mg/Day (N=26) | Placebo (N=18) | All Belumosudil (N=92)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Thalamic infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Natural death (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belumosudil 200 mg QD + Placebo (N=23) | Belumosudil 200 mg BID (Twice Daily) + Placebo (N=22) | Belumosudil 400 mg QD + Placebo (N=21) | Belumosudil 600 mg/Day (N=26) | Placebo (N=92) | All Belumosudil (N=92)
Viral upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 1 | 0 | 6
Influenza (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2
Alanine aminotransaminase (ALT) increased (Investigations) | 2 | 0 | 1 | 2 | 2 | 5
Hepatic enzyme increased (Investigations) | 2 | 1 | 0 | 2 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 2 | 5
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 4 | 1 | 1 | 1 | 6
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 2
Ligament pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 2
Meniscus injry (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 2 | 2 | 2 | 0 | 6
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 3
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT02852967/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT02852967/SAP_001.pdf